CLINICAL TRIAL: NCT01070407
Title: A Phase I Study to Assess the Safety and Immunogenicity of New Hepatitis C Virus Vaccine Candidates AdCh3NSmut and Ad6NSmut
Brief Title: A Study of a New Candidate Vaccine Against Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCV001; 2007-004259-12 (EudraCT Number); GTAC144 (Other: Gene Therapy Advisory Committee (GTAC), UK)
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C virus; HCV; Adenovirus; Vaccine
MeSH Terms: conditions — Hepatitis C; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Arm A, group 1 (Experimental): 4 volunteers
  Interventions: Biological: Ad6NSmut; AdCh3NSmut
- Arm A, group 2 (Experimental): 4 volunteers
  Interventions: Biological: Ad6NSmut; AdCh3NSmut
- Arm A, group 3 (Experimental): 5 volunteers
  Interventions: Biological: Ad6NSmut; AdCh3NSmut
- Arm B, group 5 (Experimental): 4 volunteers
  Interventions: Biological: AdCh3NSmut; Ad6NSmut
- Arm B, group 6 (Experimental): 4 volunteers
  Interventions: Biological: AdCh3NSmut; Ad6NSmut
- Arm B, group 7 (Experimental): 5 volunteers
  Interventions: Biological: AdCh3NSmut; Ad6NSmut
- Arm C, group 9 (Experimental): 5 volunteers
  Interventions: Biological: Ad6NSmut; AdCh3NSmut
- Arm C, group 10 (Experimental): 5 volunteers
  Interventions: Biological: AdCh3NSmut; Ad6NSmut
- Arm C, group 11 (Experimental): 4 volunteers
  Interventions: Biological: AdCh3NSmut; Ad6NSmut

INTERVENTIONS:
Biological: Ad6NSmut; AdCh3NSmut — 2 doses Ad6NSmut 5 x 10^8vp at weeks 0 and 4 and 1 dose AdCh3NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm A, group 1
Biological: Ad6NSmut; AdCh3NSmut — 2 doses Ad6NSmut 5 x 10^9vp at weeks 0 and 4 and 1 dose AdCh3NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm A, group 2
Biological: Ad6NSmut; AdCh3NSmut — 2 doses Ad6NSmut 2.5 x 10^10vp at weeks 0 and 4 and 1 dose AdCh3NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm A, group 3
Biological: AdCh3NSmut; Ad6NSmut — 2 doses AdCh3NSmut 5 x 10^8vp at weeks 0 and 4 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm B, group 5
Biological: AdCh3NSmut; Ad6NSmut — 2 doses AdCh3NSmut 5 x 10^9vp at weeks 0 and 4 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm B, group 6
Biological: AdCh3NSmut; Ad6NSmut — 2 doses AdCh3NSmut 2.5 x 10^10vp at weeks 0 and 4 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 24.
  Arms: Arm B, group 7
Biological: Ad6NSmut; AdCh3NSmut — 1 dose Ad6NSmut 2.5 x 10^10vp at week 0 and 1 dose AdCh3NSmut 2.5 x 10^10vp at week 8.
  Arms: Arm C, group 9
Biological: AdCh3NSmut; Ad6NSmut — 1 dose AdCh3NSmut 2.5 x 10^10vp at week 0 and 1 dose Ad6NSmut 2.5 x 10^10vp at week 8.
  Arms: Arm C, group 10
Biological: AdCh3NSmut; Ad6NSmut — 1 dose AdCh3NSmut 7.5 x 10^10vp at week 0 and 1 dose Ad6NSmut 7.5 x 10^10vp at week 8.
  Arms: Arm C, group 11

SUMMARY:
HCV001 is a Phase I study to ascertain the safety and immunogenicity of a novel vaccine against Hepatitis C virus (HCV). The vaccine is based on the sequential delivery, by intramuscular route, of two different adenoviral vectors, of human and chimpanzee origin respectively, bearing the same genetic information for HCV antigens (NS region).

The two recombinant vectors, called Ad6NSmut and AdCh3NSmut, are weakened and unable to multiply within the body; they are designed to induce an immune response against HCV proteins. Although Ad6NSmut and AdCh3NSmut have never been given to humans before this trial, promising results have been obtained in non-human studies.

The HCV001 study is designed to explore different prime-boost regimes concerning dose, order and interval of administration of Ad6NSmut and AdCh3NSmut.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 50 years (inclusive)
* Resident in or near the trial sites for the duration of the vaccination study
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective barrier contraception during the study and a negative pregnancy test on the day(s) of vaccination
* For men to use barrier contraception until three months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant simian or human adenoviral vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., Kathon
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for HIV (antibodies to HIV) at screening
* Seropositive for hepatitis C virus (antibodies to HCV) at screening
* Seropositive for simian adenovirus 3 (antibodies to AdCh3) at titres >200, at screening
* Seropositive for human adenovirus 6 (antibodies to Ad6) at titres >200, at screening
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol
* Individuals who have had a temperature >38°C in the 3 days preceding vaccination.
* Vulnerable subjects (according to the ICH E6 GCP)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety of AdCh3NSmut and Ad6NSmut, when administered in a prime/boost regimen to healthy volunteers. The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events. | Different time points depending on the study groups with a 6-months follow-up after last vaccination for all groups

SECONDARY OUTCOMES:
To assess the immunogenicity of AdCh3NSmut and Ad6NSmut, when administered in prime/boost regimen to healthy volunteers. The specific endpoint of cellular immune response will be collected via IFNγ ELIspot assay and other exploratory immunological tests. | Different time points depending on the study groups with a 6-months follow-up after last vaccination for all groups

CONTACTS AND LOCATIONS:
Overall Officials: Paul Klenerman, Professor, Study Chair — University of Oxford, UK; David Adams, Professor, Principal Investigator — University of Birmingham
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire
  - Wellcome Clinical Research Facility, Queen Elizabeth's Hospital, University Hospital Birmingham NHS Foundation Trust, Birmingham, West Midlands

REFERENCES:
- [Derived] Alsaleh G, Panse I, Swadling L, Zhang H, Richter FC, Meyer A, Lord J, Barnes E, Klenerman P, Green C, Simon AK. Autophagy in T cells from aged donors is maintained by spermidine and correlates with function and vaccine responses. Elife. 2020 Dec 15;9:e57950. doi: 10.7554/eLife.57950. PMID 33317695
- See also: HCV001 Study sponsor web site — http://www.okairos.com